CLINICAL TRIAL: NCT06151769
Title: The Effect of Topical Pomegranate Seed Oil on Prevention and Progression of Control Pressure Ulcers in Intensive Care Patients
Brief Title: The Effect Pomegranate Seed Oil Prevention and Progression Pressure Ulcers in Intensive Care Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Handan Topan, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ErciyesUnı23
Record Dates: First submitted 2023-11-14; First posted 2023-11-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; Pomegranate Seed Oil; Intensive Care
MeSH Terms: conditions — Pressure Ulcer | interventions — Sesame Oil

STUDY DESIGN:
Intervention Model Description: Pomegranate seed oil: Pomegranate seed oil will be applied to the sacrum and heels twice a day between 09.00-21.00 without pressing. This process will continue for six days.
  Sesame oil: Sesame oil will be applied to the sacrum and heels twice a day between 09.00-21.00 without pressing. This process will continue for six days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pomegranate seed oil (Experimental): In addition to the routine care of patients, pomegranate seed oil will be applied to the sacrum and heels twice a day between 09.00-21.00 without pressing. 1.5 cc will be applied to the back of the sacrum and 1 cc to each heel, using circular movements without pressure for approximately 5 seconds. It will be waited for 2-3 minutes for the body to absorb the oil, then it will be touched and removed with a napkin without any rubbing movements. The application will be applied for 6 days.
  Interventions: Other: topical pomegranate seed oil
- Sesame oil (Active Comparator): In addition to the routine care of patients, Sesame oil will be applied to the sacrum and heels twice a day between 09.00-21.00 without pressing. 1.5 cc will be applied to the back of the sacrum and 1 cc to each heel, using circular movements without pressure for approximately 5 seconds. It will be waited for 2-3 minutes for the body to absorb the oil, then it will be touched and removed with a napkin without any rubbing movements. The application will be applied for 6 days.
  Interventions: Other: Sesame oil
- Control group (No Intervention): Patients will not be interfered with in their routine care. Patient monitoring will be done every afternoon for 6 days.

INTERVENTIONS:
Other: topical pomegranate seed oil — Intervention groups: In addition to the routine care of the patients, Pomegranate seed oil will be applied to the sacrum and heels twice a day between 09.00-21.00 without pressing. 1.5 cc will be applied to the back of the sacrum and 1 cc to each heel, using circular movements without pressure for approximately 5 seconds. It will be waited for 2-3 minutes for the body to absorb the oil, then it will be touched and removed with a napkin without any rubbing movements. The application will be applied for 6 days. The patient follow-up form will be completed by the researcher every day at 12:00 noon. Again, on the 6th day of the application, evaluation surveys with the Braden risk assessment scale will be conducted by the researcher.
  Arms: Pomegranate seed oil
Other: Sesame oil — Sesame oil
  Arms: Sesame oil

SUMMARY:
Pressure sores are an important health problem that can be seen at any age and in any environment where care is provided, especially in intensive care units. It is a problem that can frequently develop, especially in people who are bedridden for long periods of time and who have acute or chronic diseases. While the incidence of pressure ulcers in hospitals is 10-23%, this rate has been reported to be 8.1%-41% in intensive care units. In Turkey, the incidence of pressure ulcers in patients receiving mechanical ventilation treatment for at least 24 hours was found to be 17% and 15.5% in intensive care units.

It is an important problem that requires long-term care and treatment after the development of a pressure sore, prolongs the duration of hospitalization, has high treatment and care costs, and increases morbidity. In a systematic review, it was stated that pressure ulcer treatment, in addition to normal treatment, increased the per capita cost of care between € 2.65 and € 87.57 per day.The care provided due to developing pressure sores increases the burden on healthcare professionals and makes it difficult to achieve the desired quality of care.It also brings an extra financial burden to care institutions.Studies have found that pressure ulcer development increases the cost of nursing care. Pressure sores also cause pain, infection, etc. in patients. It leads to the development of serious problems, deterioration in comfort and a significant decrease in the quality of life. The use of complementary medicines, including medicinal plants, has long been recommended in this regard.

The latest approaches in medicine recommend its use in the prevention and treatment of diseases due to its fewer side effects, and it is welcomed by patients. Assessment and care of the skin is important in preventing pressure sores. Pomegranate seed oil is very rich in conjugated fatty acids (linoleic and linolenic fatty acids). Although the effectiveness of pomegranate seed oil has been investigated in many subjects, there is no study examining its effectiveness in preventing and healing wound development. The aim of this study is to determine the application of topical pomegranate seed oil. To examine its effect on pressure sore development and progression. To determine the effect of topical pomegranate seed application on the prevention and progression of pressure sores. It will be conducted as a randomized controlled experimental study.

DETAILED DESCRIPTION:
Pressure sores are an important health problem that can be seen at any age and in any environment where care is provided, especially in intensive care units. It is a problem that can frequently develop especially in people who are bedridden for long periods of time and have acute or chronic diseases. While the incidence of pressure ulcers in hospitals is 10-23%, this rate has been reported to be 8.1%-41% in intensive care units. In Turkey, the incidence of pressure ulcers in patients receiving mechanical ventilation treatment for at least 24 hours was found to be 17% and 15.5% in intensive care units.

It is an important problem that requires long-term care and treatment after the development of a pressure sore, prolongs the duration of hospitalization, has high treatment and care costs, and increases morbidity. In a systematic review , it was stated that pressure sore treatment, in addition to normal treatment, increased the per capita cost of care between 2.65 € and 87.57 € per day. According to data published in the National Pressure Ulcer Advisory Panel (NPUAP) in 2016, it has been reported that the frequency of pressure ulcers in the United States is between 1.3-3 million and its annual cost is around 2.2-3.6 billion dollars. When the situation in pressure sores in our country is examined, it was determined that the average number of patients with pressure sores annually is 2.5 million and the annual cost of these patients to the country is 11.5 billion dollars.

The care provided due to developing pressure sores increases the burden of healthcare professionals and makes it difficult to achieve the desired quality of care. It also brings an extra financial burden to care institutions. Studies have found that pressure ulcer development increases the cost of nursing care.

Pressure sores also cause pain, infection, etc. in patients. It leads to the development of serious problems, deterioration in comfort and a significant decrease in the quality of life. To prevent all this, in recent years, various initiatives have been undertaken in clinical areas to prevent pressure sores and heal wounds, mainly based on the application of evidence-based guidelines. According to studies, it has been determined that different methods are used for the prevention and healing of pressure sores. In experimental or quasi-experimental studies conducted according to different methods, it was found that the development of pressure sores was not affected and in other studies it was found that it did not provide an effective change in prevalence but reduced the incidence. A study on the prevention of pressure sores, pressure-relieving mattresses and planned repositioning, anodal and cathodal-anodal electrical stimulation in category II-IV pressure sores, chronic The effects of negative pressure vacuum-assisted closure technology on the rapid healing of wounds were examined. Again, such as the effect of laser treatment on angiography, fibrogenic factors and cytokine concentrations during the healing process of pressure sores and stem cell therapy in skin wound healing methods were used. However, no definitive method to treat and prevent pressure sores has been discovered so far.

The use of complementary medicines, including medicinal plants, has long been recommended in this regard. Recent approaches in medicine recommend its use in the prevention and treatment of diseases because it has fewer side effects, and it is welcomed by patients. In a study examining the effect of olive oil on preventing pressure sores in bedridden patients, it was determined that the use of olive oil could be an effective method.

Assessment and care of the skin is important in preventing pressure sores. Dry skin is very effective in the development of pressure sores. In another study, aloe vera gel was applied to patients at risk of developing pressure sores in orthopedic clinics. No symptoms such as increased temperature, redness or swelling were observed in the areas where aloe vera gel was applied. Therefore, it can be applied to prevent pressure sores. Smooth skin is more resistant to external pressures.

Pomegranate seed oil is very rich in conjugated fatty acids (linoleic and linolenic fatty acids). It is reported that pomegranate seed oil is effective in preventing prostate and skin cancer and reducing lipid levels in the liver. Pomegranate seed oil, which has a very high vitamin E content, is also rich in antioxidant polyphenols. In a study conducted with vitamin E, it was found to be effective in oral mucositis preventive and therapeutic oral care practices.

In addition to these effects, pomegranate seed oil is one of the rare products that contain conjugated fatty acids. In a randomized controlled study examining the effect of pomegranate seed oil supplementation on Glucose transporter type 4 (GLUT-4) gene expression and glycemic control in obese people with type 2 diabetes, it was found to significantly increase Glucose transporter type 4 (GLUT-4) gene expression . In a study examining the effect of pomegranate seed oil on serum Tumor necrosis factor (TNF-α) level in dyslipidemic patients, it was found that orally administered pomegranate seed oil did not affect serum Tumor necrosis factor (TNF-α) level in patients with dyslipidemia. In another study examining the effect of pomegranate seed oil on hyperlipidemic subjects, it was found that oral pomegranate seed oil given for 4 weeks had a positive effect on the lipid levels of the patients. As can be seen, although the effectiveness of pomegranate seed oil has been investigated in many subjects in the literature review, there is no study examining its effectiveness in preventing and healing wound development.

The aim of this study is to examine the effect of topical pomegranate seed oil application on pressure ulcer development and progression.

ELIGIBILITY:
Inclusion Criteria:

* Without skin disease
* Those within the first 24 hours of admission to the intensive care clinic,
* Those with medium, high and very high risk according to the Braden risk assessment scale
* Patients without malnutrition according to CONUT score
* Those with hemoglobin level of 8 and above
* Patients who will stay in intensive care for 6 days or more
* Those with a BMI of 35 and below
* Those whose oxygen saturation is 90 and above

Exclusion Criteria:

* Those who do not allow themselves or their first degree relatives to participate in the study,
* Those with pressure sores during hospitalization,
* Those with severe edema (+4 and above),
* Those with albumin 2 and below
* Those with prealbumin 10 and below,
* Those who have a known allergy to any skin care product,
* Patients with contraindications due to brain death, cardiac arrest, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-02-18 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Nutritional Status Control (CONUT score) | first 1 day
  Parameters Normal Light Moderate Severe Serum albümin (g/dl) ≥3.5 3.0-3.49 2.5-2.9 <2.5 Score 0 2 4 6 Total lymphocyte (count/mm3) ≥1600 1200-1599 800-1199 <100 Score 0 1 2 3 Total cholesterol (mg/dl) ≥180 140-180 100-139 <100 Score 0 1 2 3 CONUT score 0-1 2-4 5-8 9-12 Assessment
Braden Risk Assessment Scale | six days
  These risk factors are evaluated by nurses and given a score between 6-23. The Braden pressure sore risk assessment scale measures the risk of pressure sores based on total scoring. 6-9 points: Very high risk, 10-12 points: High risk, 13-14 points: Medium risk
Ramsay Sedation Scale | First 1 day
  1. Awake and anxious, agitated or restless
  2. Awake, cooperative, accepting ventilation, oriented, calm
  3. Awake, only responding to commands
  4. Sleepy, has a lively/energetic response to light glabellar tapping or loud noise
  5. Sleepy, has a dull/sluggish response to light glabellar tapping or loud noise, but no response to painful sleep
  6. Sleepy, no response to light glabellar beat or loud sound
Patient Follow-up Form | six days
  It was created to record the skin evaluation of patients in the intervention and control groups before daily care, and to record blood pressure, respiratory rate, pulse, fever and saturation parameters before the application. Since blood values are checked every day in the intensive care unit, no extra blood will be taken.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Handan Topan, Kayseri
  - Handan, Kayseri

IPD SHARING:
Plan to Share IPD: No